CLINICAL TRIAL: NCT00630903
Title: Prospective, Randomized Multicentic to Compare PUVA+IFN Alpha 2a vs PUVA Alone in Mycosis Fungoides Stages Ia, Ib or IIa.
Brief Title: PUVA Versus PUVA + IFN Alpha 2a in Mycosis Fungoides
Acronym: MF99
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: Madrilenian Group of Cutaneous Lymphomas (Other)
Responsible Party: Dr F Vanaclocha Sebastián, Servicio de Dermatología. Hospital 12 de Octubre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MF99
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-02

CONDITIONS: Cutaneous T-Cell Lymphoma (Mycosis Fungoides)
MeSH Terms: conditions — Mycosis Fungoides | interventions — Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): 8-MOP + UVA x 24 weeks
  Interventions: Drug: PUVA (8-MOP + UVA)
- B (Active Comparator): IFN alone, 2 weeks, 8-MOP + UVA irradiation + IFN, 22 weeks
  Interventions: Drug: PUVA (8MOP + UVA) + IFN

INTERVENTIONS:
Drug: PUVA (8MOP + UVA) + IFN — Weeks 3-24: 8.MOP: 0.6 MG/K, 3 times a week, 2 hours pre UVA irradiation (1-2 jul/cm2 according to phototype, increasing until 10 Jul/cm2, if tolerated) IFN: week1: 3, 6 and 9 MU (Mon, Wed, Fry). Weeks 2-24: 9MU 3 times a week)
  Arms: B
Drug: PUVA (8-MOP + UVA) — Weeks 1-24: 8.MOP: 0.6 MG/K, 3 times a week, 2 hours pre UVA irradiation (1-2 jul/cm2 according to phototype, increasing until 10 Jul/cm2, if tolerated)
  Arms: A

SUMMARY:
The purpose of this study is to determine if combination of PUVA with interferon alpha is better than PUVA alone to treat mycosis fungoides stage Ia Ib or IIa.

ELIGIBILITY:
Inclusion Criteria:

* Mycosis fungoides Stage Ia Ib IIa
* Written informed consent
* 18-70 y.o., both sex
* No concomitant systemic disease

Exclusion Criteria:

* Pregnant or lactating women
* Fertile women not accepting contraception
* Medical history of melanoma or non melanoma skin cancer
* Concomitant infections
* Immunodeficiency states
* Previous Heart disease
* Respiratory insufficiency
* Chronic RRenal insufficiency
* Chronic hepatopathy
* Epilepsy
* Depression
* Leucocytes <3000 or neutrophiles <1000 or thrombocytes <100000 or hemoglobin <12 gr/dL or ANA <1/80
* Treatment with systemic steroids
* Altered thyroid hormones
* Previous resistance to PUVA and/or IFN
* Hypersensitivity to IFN
* Patients under treatment with teophiline and/or dicumarol
* Previous total skin electron beam
* Wash up period less than 3 month for IFN and /or PUVA
* Wash up period less than 1 month for topical treatments

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-01; Primary Completion 2003-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PUVA vs PUVA + IFN | Weeks 4, 8, 12, 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Vanaclocha Sebastián, MD, Principal Investigator — Hospital 12 de Octubre; Jesús Fernández Herrera, MD, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (9):
- Spain (9):
  - Hospital Príncipe de Asturias., Alcalá de Henares, Madrid
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital de la Princess, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Gómez Ulla, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956